CLINICAL TRIAL: NCT04464317
Title: Vocal Cord Impairment and Dysphagia in Cardiac Surgery
Brief Title: Dysphagia and Vocal Cord Injury Following Cardiac Surgery
Status: Withdrawn | Type: Observational
Why Stopped: Observational only, no subjects enrolled
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB202001240
Record Dates: First submitted 2020-06-30; First posted 2020-07-09 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Dysphagia; Cardiovascular Diseases
MeSH Terms: conditions — Deglutition Disorders; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient who has had cardiovascular surgery: Undergone an elective, urgent, and/or emergent cardiovascular surgery via endovascular or open (sternotomy and/or extended thoracotomy) technique at the University of Florida Health.

SUMMARY:
Aiming to determine the incidence and contributing risk factors of vocal fold mobility impairment (VFMI) and dysphagia in postoperative cardiovascular patients and evaluate the impact of VFMI on health-related outcomes.

DETAILED DESCRIPTION:
This is a retrospective study to determine:

1. the incidence and contributing risk factors of vocal fold mobility impairment (VFMI) and dysphagia in postoperative cardiovascular patients
2. evaluate the impact of VFMI on health-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All cardiac surgery patients January 2010-April 2020 at Shands Hospital
* Patients aged between 18 and 90 years
* Undergone an elective, urgent, and/or emergent cardiovascular surgery via endovascular or open (sternotomy and/or extended thoracotomy) technique at the University of Florida Health.

Exclusion Criteria:

* Under 18 years old or over 90 years old

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone an elective, urgent, and/or emergent cardiovascular surgery via endovascular or open (sternotomy and/or extended thoracotomy) technique at the University of Florida Health.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2023-06-13 (Estimated); Study Completion 2023-06-13 (Actual)

PRIMARY OUTCOMES:
Incidence of vocal fold mobility impairment (VFMI) and dysphagia in postoperative cardiovascular patients | January 2010-June 2020
  Data analyses will be conducted using commercially available statistical software, SPSS and only de-identified data will be used during data analysis. We will pull data from the files in order to determine how often the patients have vocal fold mobility impairment and/or dysphagia following surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jeng, MD, Principal Investigator — University of Florida

IPD SHARING:
Plan to Share IPD: No
none at this time